CLINICAL TRIAL: NCT04792333
Title: A Phase I Study to Compare Pharmacokinetic Parameters of Firibastat and Its Metabolites (EC33 and QGC515) in Healthy Subjects Versus End Stage Renal Disease (ESRD) Patients After a Single Oral Administration of Firibastat 500 mg
Brief Title: Pharmacokinetics in End Stage Renal Disease Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Quantum Genomics SA (Industry)
Collaborators: Eurofins Optimed (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: QGC001-1QG4; 2019-001817-18 (EudraCT Number)
Record Dates: First submitted 2019-12-26; First posted 2021-03-10 (Actual); Last update posted 2021-03-10 (Actual); Status verified 2021-03

CONDITIONS: Healthy Volunteers; Renal Failure
MeSH Terms: conditions — Renal Insufficiency | interventions — firibastat

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment (Experimental): 500 mg (2 capsules of 250 mg)
  Interventions: Drug: firibastat

INTERVENTIONS:
Drug: firibastat — Single oral dose of 500 mg administration on Day 1
  Other Names: QGC001

SUMMARY:
The study is a multicentre, open label, phase I, two arms study to compare pharmacokinetic of firibastat after a single oral dose of firibastat 500 mg in fourteen healthy male volunteers and in fourteen End Stage Renal Disease (ESRD) patients not yet in dialysis.

DETAILED DESCRIPTION:
It is planned to enroll a total of 28 subjects to receive a single oral dose of investigational medicinal product (IMP): 14 ESRD patients will be enrolled in three Hungarian centres (1st arm) and 14 Healthy volunteers will be enrolled by Eurofins Optimed in Gières, France (2nd arm).

Subjects will be screened for eligibility to participate in the study up to 21 days prior to the first administration. For both arm, subjects will be admitted into the Clinical Research Unit (CRU) on Day -3. On the morning of Day 1, subjects will receive a single 500 mg oral dose of firibastat following an overnight fast (i.e., at least 10 hours). Subjects will be confined to the CRU until discharge on Day 3 with PK blood sample draws for measurement of firibastat and its main metabolites being taken throughout the confinement.

A follow-up post study visit will occur on Day 10 post-dose to ensure the ongoing wellbeing of the subjects.

ELIGIBILITY:
Inclusion Criteria:

* Male subjects, aged 18 to 55 years inclusive;
* Non-smoker subject or smoker of not more than 5 cigarettes a day;

Exclusion Criteria:

* Positive Hepatitis B surface (HBs) antigen or anti Hepatitis C Virus (HCV) antibody, or positive results for Human Immunodeficiency Virus (HIV) 1 or 2 tests);
* History or presence of drug or alcohol abuse (alcohol consumption > 40 grams/day);

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2019-09-17 (Actual); Primary Completion 2020-07-10 (Actual); Study Completion 2020-07-10 (Actual)

PRIMARY OUTCOMES:
Firibastat and metabolites Concentrations | Day 1 to Day 3
  The plasma concentration data for firibastat (QGC001), EC33 and QGC515, will be analysed at each time measurement (predose, 0, 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 16, 24, 36, 48 hours post-dose)

SECONDARY OUTCOMES:
Systolic and Diastolic Blood Pressure (mmHg) | Day 1 to Day 3
  Systolic and Diastolic blood pressure
Heart Rate (bpm) | Day 1 to Day 3
  number of beats per minute
Hematology blood sample laboratory tests aggregated as number of patients outside ranges | Day 1 to Day 3
  Hemoglobin, Hematocrit, MCH, MCHC, MCV, MPV, RBC (erythrocytes), WBC (Leucocytes), Differential Count (Basophils, Eosinophils, Lymphocytes, Monocytes, Neutrophils, Large Unstained cells), Platelets.
Biochemistry blood sample laboratory tests aggregated as number of patients outside ranges | Day 1 to Day 3
  Albumin, Alkaline Phosphatase, ALT, Amylase, AST, Bicarbonate, Bilirubin (direct, indirect and total), Calcium, Chloride, Cholesterol, Creatinine Kinase, Creatinine, gammaGT, HDLcholesterol, LDH, LDL - cholesterol, Lipase, Magnesium, Phosphate, Potassium, Protein total, Sodium, Triglycerides, Urea, Uric Acid, Glucose.
Hemostasis blood sample laboratory tests aggregated as number of patients outside ranges | Day 1 to Day 3
  INR, PT, aPTT
Urinalysis tests aggregated as number of patients outside ranges | Day 1 to Day 3
  pH, ketone bodies, proteins, glucose, occult blood, blood leukocytes, nitrite, bilirubin, urobilinogen, density.

CONTACTS AND LOCATIONS:
Overall Officials: Yves DONAZZOLO, MD, Principal Investigator — Eurofins Optimed
Locations (1):
- Eurofins Optimed, Gières, France

IPD SHARING:
Plan to Share IPD: No